CLINICAL TRIAL: NCT06888674
Title: Clinical Study to Evaluate the Safety and Efficacy of Personalized Tumor Neoantigen MRNA Therapy Combined with PD-1 Antibody and Chemotherapy As Adjuvant Treatment for Postoperative Pancreatic Cancer.
Brief Title: Personalized Tumor Neoantigen MRNA Therapy Adjuvant Treatment for Postoperative Pancreatic Cancer.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CISPD-11
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer Resectable
MeSH Terms: interventions — Gemcitabine; Capecitabine; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Chemotherapy-Tolerant Patients) (Experimental): Postoperative evaluation will be conducted within 4-12 weeks after surgery, and patients without recurrence will be enrolled. For patients who are chemotherapy-tolerant (evaluated by investigators), adjuvant therapy is to commence within 6-12 weeks postoperatively, with the first day of treatment (D1) defined as the date of initial postoperative intervention. Postoperative treatment follows the:
  1.Gemcitabine + Capecitabine (GC) regimen+ Sintilimab: Gemcitabine: 1000 mg/m², intravenously on D1 and D8;Capecitabine: 1650-2000 mg/(m²·day), divided into two daily oral doses from D1 to D14；Sintilimab (200 mg); Q3W for 8 cycles.2.Personalized mRNA injection (100 μg subcutaneously, Q3W) administered from D22±3.
  On Day 43 ±3 days: The second efficacy assessment will be performed. Patients without disease progression will continue treatment. Patients with disease progression will transition to a second-line chemotherapy regimen (decided by investigators) combined with mRNA and Sintilimab.
  Interventions: Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection; Drug: Gemcitabine + Capecitabine; Drug: Sintilimab injection
- Arm B (Chemotherapy-Intolerant or Chemotherapy-Declined Patients) (Experimental): Postoperative evaluation will be conducted within 4-12 weeks after surgery, and patients without recurrence will be enrolled. For patients who are Chemotherapy-Intolerant or Chemotherapy-Declined, postoperative treatment consists of Sintilimab (200 mg via intravenous infusion) administered Q3W for 8 cycles. On Day 22 ± 3 days, patients will initiate treatment with personalized mRNA injection at a dose of 100 μg administered subcutaneously Q3W, for a maximum of 9 doses.
  On Day 43 ±3 days: The second efficacy assessment will be performed. Patients without disease progression will continue treatment. Patients with disease progression will transition to a second-line chemotherapy regimen (decided by investigators) combined with personalized mRNA injection (100 μg subcutaneously,Q3W) and Sintilimab (200 mg via intravenous infusion, Q3W).
  Interventions: Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection; Drug: Sintilimab injection

INTERVENTIONS:
Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection — The individualized anti-tumor new antigen iNeo-Vac-R01 injection was commissioned by Hangzhou Neoantigen Therapeutics Co., Ltd., and all patients were admitted into the therapeutic intervention group. According to the results of previous non-clinical studies, the individualized mRNA injection of 100 μ g was a tolerable dose.
Drug: Gemcitabine + Capecitabine — Gemcitabine: 1000 mg/m², administered intravenously over 30 minutes on Day 1 and Day 8; Capecitabine: 1650-2000 mg/(m²·day), divided into two daily oral doses from Day 1 to Day 14.
  Treatment cycles repeat every 3 weeks for 8 cycles, with the actual number of cycles determined by the investigator based on comprehensive evaluation of the patient's physical status, disease progression, and adverse reactions.
  Arms: Arm A (Chemotherapy-Tolerant Patients)
Drug: Sintilimab injection — Sintilimab Injection, 200mg, intravenous infusion, every 3 weeks

SUMMARY:
This study is a single-center, open-label clinical study to evaluate the feasibility and safety of personalized tumor neoantigen mRNA therapy (iNeo-Vac-R01) in combination with PD-1 antibody and standard chemotherapy regimen as adjuvant treatment for postoperative resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-Screening Phase Inclusion Criteria (for Radical Surgery and Vaccine Preparation):

   * Subjects meeting all of the following criteria will enter the pre-screening phase for radical surgery and vaccine preparation:
   * Voluntarily sign the informed consent form (ICF);
   * Age ≥18 years, regardless of gender;
   * Diagnosed with resectable pancreatic cancer as assessed per the 2024 NCCN Clinical Practice Guidelines and willing to undergo radical surgery;
   * ECOG Performance Status score of 0 or 1;
   * Ability to obtain sufficient fresh tumor tissue samples for whole-exome sequencing (WES) and transcriptome sequencing analysis;
   * Normal function of major organs (heart, liver, kidneys):
   * Liver function: Total bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN;
   * Renal function: Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault formula);
   * Cardiac function: LVEF ≥50% by echocardiography;
   * Contraception agreement: Fertile males and females of childbearing potential must agree to use effective contraception from signing the ICF until 6 months after the last dose of study treatment. Females of childbearing potential include premenopausal women and women ≤2 years postmenopausal;
   * Ability to comply with the study protocol and follow-up procedures.
2. Formal Screening Phase Inclusion Criteria (for Study Treatment Initiation):

   * Subjects meeting all of the following criteria will enter the formal screening phase for study treatment:
   * Voluntarily sign the informed consent form (ICF);
   * Age ≥18 years, regardless of gender;
   * Histologically confirmed pancreatic ductal adenocarcinoma (PDAC) post-surgery;
   * Completion of radical resection (R0 or R1) with no evidence of metastatic disease, malignant ascites, or pleural effusion on imaging 4-12 weeks postoperatively;
   * ECOG Performance Status score:Cohort A: 0 or 1;Cohort B: 0-2;
   * Normal function of major organs (heart, liver, kidneys):
   * Contraception agreement: Same as pre-screening criteria;
   * Ability to comply with the study protocol and follow-up procedures.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

* Serum CA 19-9 level >180 U/mL within 21 days prior to initiating standard postoperative adjuvant therapy;
* History of bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation;
* Concurrent immunosuppressive therapy, defined as regular use of immunosuppressive agents within 4 weeks prior to screening or during the study, including but not limited to:

  1. Severe asthma requiring systemic corticosteroids (≥10 mg/day prednisone equivalent);
  2. Active autoimmune disease or immunodeficiency (e.g., rheumatoid arthritis, systemic lupus erythematosus);
  3. History of primary immunodeficiency;
  4. Exceptions: Type 1 diabetes, autoimmune hypothyroidism managed with hormone replacement, vitiligo, or psoriasis not requiring systemic therapy;
* Active bacterial/fungal infections requiring systemic treatment, or active/latent tuberculosis (confirmed by interferon-gamma release assay or tuberculin skin test);
* Active viral infections:

  1. HIV antibody-positive;
  2. Syphilis (TP antibody-positive with RPR/TRUST confirmation);
  3. Active hepatitis C (HCV RNA-positive);
  4. Active hepatitis B (HBsAg-positive and HBV DNA ≥2000 IU/mL);
* Acute viral infections:

  1. Herpesvirus infection (unless resolved with crusting >4 weeks prior);
  2. Respiratory viral infection (unless resolved >4 weeks prior);
* Uncontrolled comorbidities:

  1. Symptomatic congestive heart failure (NYHA Class III/IV);
  2. Unstable angina or arrhythmia requiring treatment;
  3. Severe coronary/cerebrovascular disease (e.g., myocardial infarction within 6 months);
  4. Other conditions deemed exclusionary by the investigator;
* History of drug abuse, psychiatric disorders, or psychosocial factors impairing informed consent or protocol compliance;
* History of severe hypersensitivity to vaccines, biologics, or any component of the study drug;
* Pregnancy or lactation;
* Other conditions judged by the investigator to preclude safe participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurence and frequence of AE and SAE | Up to 2 years
  Occurence and frequence of Adverse Event (AE) and Serious Adverse Event (SAE) (NCI CTCAE 5.0)

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 2 years
  Defined as the time from the date of surgery to the first occurrence of disease recurrence or death from any cause (whichever occurs first). Tumor recurrence is defined as the development of one or more new lesions, which may be local (at the primary site), regional (in adjacent lymph nodes or tissues), or distant (metastatic lesions remote from the original resection site).
Recurrence-Free Survival Rate (RFS%) | Up to 3 years
  The proportion of patients free from disease recurrence or death (whichever occurs first) at 12 months, 24 months, and 36 months following surgery.
Overall Survival (OS) | Up to 4 years
  Defined as the time from the date of surgery to death from any cause.
Overall Survival Rate (OS%) | Up to 3 years
  The proportion of patients surviving at 12 months, 24 months, and 36 months following surgery.
Efficacy Evaluation Metrics for Patients with Recurrence: Objective Response Rate (ORR) | Up to 3 years
  The proportion of patients achieving a partial response (PR) or complete response (CR) in tumor lesions, as defined by RECIST 1.1 criteria.
Efficacy Evaluation Metrics for Patients with Recurrence: Disease Control Rate (DCR) | Up to 3 years
  The proportion of patients achieving PR, CR, or stable disease (SD) in tumor lesions.
Efficacy Evaluation Metrics for Patients with Recurrence: Progression-Free Survival (PFS) | Up to 3 years
  Defined as the time from the date of initiating first-line chemotherapy to the first occurrence of disease progression or death from any cause (whichever occurs first).
Efficacy Evaluation Metrics for Patients with Recurrence: Progression-Free Survival Rate (PFS%) | Up to 3 years
  The proportion of patients free from disease progression or death (whichever occurs first) at 12, 24, and 36 months.
Efficacy Evaluation Metrics for Patients with Recurrence: Overall Survival (OS) | Up to 4 years
  Defined as the time from the date of initiating first-line chemotherapy to death from any cause.
Efficacy Evaluation Metrics for Patients with Recurrence: Overall Survival Rate (OS%) | Up to 3 years
  The proportion of patients surviving at 12, 24, and 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No